CLINICAL TRIAL: NCT05237206
Title: A Phase 1, First-in-Human, Open-label Single Agent Study of SUPLEXA Therapeutic Cells in Patients With Metastatic Solid Tumours and Haematologic Malignancies
Brief Title: Study of SUPLEXA in Patients With Metastatic Solid Tumours and Haematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alloplex Biotherapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUPLEXA-101
Record Dates: First submitted 2022-02-01; First posted 2022-02-14 (Actual); Results first posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-08

CONDITIONS: Oncology
Keywords: autologous therapy; cellular therapy; T cell; NK-T cell; gamma delta T cell; CTL; PBMC-derived effector cells; NK cells
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: non-comparative, open-label, basket-design study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SUPLEXA (Experimental): autologous cellular therapy comprised predominantly of NK, NK-T, and T cells stored in cryogenic media
  Interventions: Biological: SUPLEXA

INTERVENTIONS:
Biological: SUPLEXA — PBMC-derived autologous cellular therapy derived through an ex vivo activation procedure, resulting in a cell mixture comprised predominantly of NK, NK-T, and T cells stored in cryogenic media.

SUMMARY:
This Phase 1, first-in-human (FIH), open-label study is designed to assess the safety, tolerability, and preliminary clinical efficacy of repeated intravenous (IV) infusions of SUPLEXA monotherapy in subjects with measurable metastatic solid tumours and haematologic malignancies

DETAILED DESCRIPTION:
This is a FIH Phase 1, non-comparative, open-label, basket-design study. The study will consist of 2 cohorts:

* Solid tumours cohort
* Haematologic malignancies cohort:

Subjects must fulfill entry criteria and have relapsed or refractory advanced malignancy for which no standard therapy exists.

An Data Safety Monitoring Committee (DSMB) will provide oversight of the study and will monitor safety on a regular basis throughout the study to make recommendations on any modifications.

The study will be comprised of 3 periods. Screening, Treatment and Follow-up.

All eligible subjects will receive minimally 3 weekly dosing of SUPLEXA. Subjects will be monitored closely at the clinic after each weekly infusion.

After completion of the first 3 weekly SUPLEXA the treatment period of SUPLEXA may be extended to every 2 weeks until all SUPLEXA is depleted.

ELIGIBILITY:
Inclusion Criteria:

* Age

  1. Adult subjects at least 18 years of age at the time of signing the PICF.

     Type of Subject and Disease Characteristics Solid Tumours
  2. Histologically or cytologically confirmed diagnosis of locally advanced or metastatic solid tumour.
  3. Have 1 or more tumours measurable based on RECIST v1.1 as assessed by the local site Investigator. Radiographic scans should be obtained within 4 weeks of Screening. Lesions situated in a previously irradiated area are considered measurable if objective progression has been demonstrated following radiation to such lesions.
  4. Subjects who did not attain a durable response after receiving at least one standard/approved therapies which may include chemotherapy, targeted agents, radio-, immuno- conjugates, check point inhibitors or where there is no approved therapy. This includes subjects who attained a long-term stable disease (SD), or partial response (PR) are eligible. Long term SD subjects on a checkpoint inhibitor may continue checkpoint inhibitor (CPI) therapy.

     Haematologic malignancies
  5. Histologically or cytologically confirmed multiple myeloma, lymphoma, and chronic lymphocytic leukemia (collectively termed as haematologic malignancies for the purposes of this protocol) which has relapsed or is refractory advanced malignancy for which no curative standard therapy exists.

Exclusion Criteria:

Medical Conditions

1. Known central nervous system (CNS) metastases and/or carcinomatous meningitis.
2. Prior allogeneic transplant.
3. Diagnosis of immunodeficiency or is receiving chronic and non-physiological, systemic steroid therapy or any other form of immunosuppressive therapy.
4. Active uncontrolled bacterial, viral, or fungal infection requiring systemic therapy at screening or Day 1.
5. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating Investigator.
6. Any unresolved Grade 2 or greater reversible toxicity from a previous anticancer therapy except for alopecia or Grade 2 neuropathy.
7. Clinically significant cardiovascular disease, including any of the following:

   1. Stroke or myocardial infarction within 6 months prior to first dose in the study.
   2. Presence of unstable angina within 6 months prior to first dose in the study.
   3. Congestive heart failure of New York Heart Association Grade 2 or higher.
   4. History or presence of clinically significant ventricular arrhythmias, or conduction abnormality; presence of clinically significant atrial fibrillation and resting bradycardia.
   5. Corrected QT interval (QTcF) of >450 msec (males) or >470 msec (females) using Fridericia's correction formula.
   6. History of congenital long QT syndrome.
8. Known history of testing positive for human immunodeficiency virus (HIV), and/or positive test for Hepatitis B virus surface antigen (HBsAg) and/or positive Hep C antibody result with detectable hepatitis C virus (HCV) ribonucleic acid (RNA) indicating acute or chronic infection.
9. A serious non-malignant disease (e.g., psychiatric, substance abuse, uncontrolled intercurrent illness, etc.) that could compromise protocol objectives in the opinion of the Investigator and/or the Sponsor.
10. At high risk of developing TLS per (Cairo, 2010)). Specifically:

    1. Burkitt's lymphoma
    2. ALL with LDH > 2xULN or WBC >100 x 109 per µL.
    3. AML with WBC >100 x 109 per µL.
11. Any other condition that, in the opinion of the Investigator, would prohibit the subject from effectively participating in the study.

    Diagnostic Assessments
12. A performance status ≥2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale (solid tumours cohort) or Karnofsky performance scale of ≥60 (haematologic malignancies cohort)
13. Does not demonstrate adequate organ function as defined as an excursion beyond the acceptable limits below. All screening laboratories should be performed at screening and on the day of first administration of study therapy.
14. Prior radiotherapy within 2 weeks of start of study intervention. Subjects must have recovered from all radiation-related toxicities and not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤2 weeks of radiotherapy) to non-CNS disease.
15. Transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (CSF) (including granulocyte CSF [GCSF], granulocyte-macrophage CSF [GMCSF], or recombinant erythropoietin) within 4 weeks prior to baseline.
16. Any vaccines (live, attenuated, inactivated or research vaccines) within 30 days of dosing with study intervention (refer to Section 6.8.1 for prohibited vaccines).

    Prior/Concurrent Clinical Study Experience
17. Participation in another clinical study of an investigational agent during the 2 weeks of this study's screening.

    Other Exclusions
18. < 6 months life expectancy at the local site Investigator judgement.
19. Pregnant or breastfeeding female subjects within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Joshi, MD, Principal Investigator — Cancer Research South Australia (CRSA)
Locations (3):
- Australia (3):
  - Greenslopes Private Hospital/Gallipoli Medical Research Foundation, Brisbane, Queeensland
  - Cancer Research Sa (Crsa), Adelaide, South Australia
  - Southern Oncology Clinical Research Unit (SOCRU), Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Poster presentation at Society for Immunotherapy of Cancer by Alloplex Biotherapeutics, presenting results from this clinical trial. — https://alloplexbio.com/publications/final-safety-and-efficacy-update-of-suplexa-101-a-first-in-human-single-agent-study-of-suplexa-therapeutic-cells-in-metastatic-solid-tumors/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from CANCER RESEARCH SA, Greenslopes Private Hospital/Gallipoli Medical Research Foundation and Southern Oncology Clinical Research Unit in Australia starting April 2022 to January 2024.
Groups:
- SUPLEXA: Autologous, non-engineered cellular therapy comprised of lymphoid cells activated through a proprietary ex vivo procedure. A cryogenically stored product was prepared for all eligible participants to receive this adoptive immune cell therapy
Period: Overall Study
Arm/Group | SUPLEXA
Started | 46
Allocated to Intervention | 35
Analyzed | 35
Completed | 35
Not Completed | 11
Not completed — screen failure-did not receive treatment | 8
Not completed — did not receive treatment | 3

BASELINE CHARACTERISTICS:
Arm/Group | SUPLEXA
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: Participants]
  Australia | 35
Age of Participants [Median (Standard Deviation); unit: years] | 64 (10.1)
Ethnicity of participants [Count of Participants; unit: Participants]
  Asian | 4
  White | 31

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of SUPLEXA in Subjects With Malignant Solid Tumour and Haematologic Malignancies.
Description: Incidence of dose limiting toxicities measured by Incidence of adverse events and serious adverse events overall, by severity, by relationship to each study intervention, and those that led to discontinuation of study intervention. Note: due to patient availability, only solid tumour patients were enrolled
Time Frame: 24 months
Population: Intent to Treat Population (all participants allocated intervention) were assessed for adverse events.
Measure: Number; unit: Participants
Arm/Group | SUPLEXA
Number analyzed (Participants) | 35
Participants
  Number of Subjects reporting any Treatment Emergent Adverse Events | 25
  Numer of Subjects reporting TEAE related to study intervention | 3
  Number of Subjects with TEAE leading to discontinuation of study intervention | 2

2. Secondary Outcome: Solid Tumours Cohort: To Assess the Efficacy of SUPLEXA in Subjects With Malignant Solid Tumour as Assessed by the Investigator Based on Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 or by Changes in Tumour-derived Blood Biomarkers.
Description: Objective response rate defined as the proportion of subjects with best overall response of either a complete response (CR) or partial response (PR) measured by Time to Progression (TTP). Complete Response (CR) is defined as disappearance of all target lesions; Partial Response (PR), is defined as at least 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: 24 months
Measure: Number (95% Confidence Interval); unit: Number of participants: ORR
Arm/Group | SUPLEXA
Number analyzed (Participants) | 35
Number of participants: ORR | 3 [2 to 5]

ADVERSE EVENTS:
Time Frame: from enrollment through end of follow up, up to 24 months
Description: The adverse events were gathered in Common Terminology Criteria for Adverse Events v.5.0
Arm/Group | SUPLEXA
All-Cause Mortality (participants affected / at risk) | 1/35
Serious Adverse Events (participants affected / at risk) | 6/35
Other Adverse Events (participants affected / at risk) | 25/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SUPLEXA (N=35)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) — Information collected at study visits through patient reported outcomes; one case determined to be Grade 3 (severe)
Gasteroenteritis astroviral (Infections and infestations) | 1 (1) — Information collected at study visits through patient reported outcomes; one case determined to be Grade 3 (severe)
Ascites (Gastrointestinal disorders) | 1 (1) — Information collected at study visits through patient reported outcomes; one case determined to be Grade 3 (severe)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) — Information collected at study visits through patient reported outcomes; one case determined to be Grade 3 (severe)
Rectal Haemorrhage (Gastrointestinal disorders) | 1 (1) — Information collected at study visits through patient reported outcomes; one case determined to be Grade 4 (Life Threatening)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Information collected at study visits through patient reported outcomes; one case determined to be Grade 3 (severe)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Information collected at study visits through patient reported outcomes; one case determined to be Grade 4 (severe)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SUPLEXA (N=35)
Constipation (Gastrointestinal disorders) | 6 (6) — Information collected at study visits through patient reported outcomes; 2 determined to be Grade 1 (mild) and 4 determined to be Grade 2 (moderate
Intestinal Obstruction (Gastrointestinal disorders) | 3 (3) — Information collected at study visits through patient reported outcomes; 2 occurrences determined to be Grade 2 (moderate) and 1 occurrence determined to be Grade 3 (severe)
Nausea (Gastrointestinal disorders) | 5 (6) — Information collected at study visits through patient reported outcomes; 2 determined to be Grade 1 (mild) and 3 determined to be Grade 2 (moderate)
Vomiting (Gastrointestinal disorders) | 2 (2) — Information collected at study visits through patient reported outcomes; 2 cases determined to be Grade 1 (mild)
Fatigue (General disorders) | 8 (9) — Information collected at study visits through patient reported outcomes
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) — Information collected at study visits through patient reported outcomes; 1 case determined to be Grade 1 (mild) and 1 determined to be Grade 2 (moderate)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) — Information collected at study visits through patient reported outcomes
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (4) — Information collected at study visits through patient reported outcomes; 1 determined to be Grade 1 (mild) and 1 determined to be Grade 2 (moderate)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) — Information collected at study visits through patient reported outcomes; one determined to be Grade 1 (mild) and one determined to be Grade 2 (moderate)
Ageusia (Nervous system disorders) | 2 (2) — Information collected at study visits through patient reported outcomes; 2 cases determined to be Grade 1 (mild)
Dizziness (Nervous system disorders) | 2 (3) — Information collected at study visits through patient reported outcomes
Headache (Nervous system disorders) | 3 (3) — Information collected at study visits through patient reported outcomes; 3 cases determined to be Grade 1 (mild)
Dizziness (Nervous system disorders) | 2 (3) — Information collected at study visits through patient reported outcomes; 3 cases determined to be Grade 1 (mild)
Insomnia (Psychiatric disorders) | 2 (3) — Information collected at study visits through patient reported outcomes
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7) — Information collected at study visits through patient reported outcomes
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) — Information collected at study visits through patient reported outcomes; 2 determined to be Grade 1 (mild), 1 determined to be Grade 2 (moderate)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/06/NCT05237206/Prot_SAP_000.pdf